CLINICAL TRIAL: NCT00511524
Title: An Open Label Positron Emission Tomography (PET) Study to Investigate Brain Penetration by [11C]GW842166 in Healthy Subjects
Brief Title: An Imaging Study to Investigate the Distribution of GW842166X in the Brain.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CBA103679
Record Dates: First submitted 2007-08-02; First posted 2007-08-06 (Estimated); Last update posted 2017-08-07 (Actual); Status verified 2017-08

CONDITIONS: Pain, Inflammatory
Keywords: brain,; inflammation,; CB2,; PET; analgesia,
MeSH Terms: conditions — Pain; Inflammation; Agnosia | interventions — 2-((2,4-dichlorphenyl)amino)-N-((tetrahydro-2H-pyran-4-yl)methyl)-4-(trifluoromethyl)-5-pyrimidinecarboxamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Subjects receiving GW842166 (Experimental): Subjects will receive single oral dose of 400 milligram (mg) un-labeled GW842166X. After 2-5 hours subjects will receive [carbonyl-^11C]GW842166.
  Interventions: Drug: GW842166X; Drug: [carbonyl-^11C]GW842166

INTERVENTIONS:
Drug: GW842166X — GW842166X will available with dose strength of 100 mg capsules. Four 100mg GW842166X capsules will be used for the 400 mg oral dose of GW842166X.
Drug: [carbonyl-^11C]GW842166 — [carbonyl-^11C]GW842166 will b available as Intravenous solution.

SUMMARY:
GW842166X is being developed for the treatment and management of inflammatory pain. GW842166X is a CB2 receptor agonist and the mechanism is not fully understood, although it is thought that for the anti-inflammatory action the drug is required to cross inot the brain from the blood. This study aims to look at if the drug crosses into the brain once given orally using an imaging technique called positron emission tomography.

ELIGIBILITY:
Inclusion Criteria:

* Male aged 50 to 80yrs inclusive at the screening visit.
* subjects with negative HIV and hepatitis B and C test results within 3 months of study start.

Exclusion Criteria:

* A negative Allens test on arm to be used for arterial cannulation.
* Any contraindications to MRI scanning.
* History or presence of hepatic or renal disease.
* Previous involvement in PET or radiological investigations.
* Family history of cancer.
* History of claustrophobia
* Presence of a cardiac pacemaker or any other electronic device or ferromagnetic metal

Ages: 50 Years to 80 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2007-06-26 (Actual); Primary Completion 2007-07-04 (Actual); Study Completion 2007-07-04 (Actual)

PRIMARY OUTCOMES:
Rate at which the drug crosses from plasma to brain (ki)using images from the scan | throughout the study

SECONDARY OUTCOMES:
Safety of drug | after taking the drug pre-dose, 2hr, 4hr, 6hr, 10hr, 24hr, follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Uppsala, Sweden

REFERENCES:
- See also: Results for study CBA103679 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/CBA103679?search=study&search_terms=CBA103679#rs